CLINICAL TRIAL: NCT00480194
Title: A Non-interventional, Non-controlled, Post-marketing Study to Obtain Knowledge of the Safety of ZyComb® (Xylometazoline Hydrochloride 0.5 mg/mL and Ipratropium Bromide 0.6 mg/mL) for Symptoms of Common Cold in a Real-life OTC Setting
Brief Title: Evaluation of Safety of ZyComb® In Patients With Common Cold - ZIP 3000 (XY-005-IM)
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Nycomed
Other Study IDs: XY-005-IM
Record Dates: First submitted 2007-05-24; First posted 2007-05-30 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-02

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — xylometazoline; Ipratropium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: xylometazoline hydrochloride and ipratropium bromide (ZyComb) — Common cold in a real-life OTC setting

SUMMARY:
The objectives of the study are to obtain knowledge about the safety in use, the patients' general impression of the treatment and the pattern of use of ZyComb® in an over-the-counter (OTC) setting.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion the patient must buy ZyComb® nasal spray with the intention to start using it either the same or the next day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For inclusion the patient must buy ZyComb® nasal spray with the intention to start using it either the same or the next day. Male or female patients over 18 years of age, visiting any of the participating pharmacies are eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters